CLINICAL TRIAL: NCT00528606
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of AA4500 in the Treatment of Subjects With Dupuytren's Contracture
Brief Title: AA4500 (XIAFLEX™, Proposed Name) in the Treatment of Dupuytren's Contracture
Acronym: CORD-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUX-CC-857
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2010-10-22 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Dupuytren's Contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA4500 0.58 mg (Experimental)
  Interventions: Biological: collagenase clostridium histolyticum
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: collagenase clostridium histolyticum — Subjects could have received up to three injections of AA4500 into the cord of the affected hand. Each injection was separated by at least 30 days. Individual cords may have received up to a maximum of three injections.
  Other Names: XIAFLEX®; AA4500
  Arms: AA4500 0.58 mg
Biological: Placebo — Subjects could have received up to three injections of placebo into the cord of the affected hand. Each injection was separated by at least 30 days. Individual cords may have received up to a maximum of three injections.
  Arms: Placebo

SUMMARY:
This was a Phase 3, double-blind, randomized, placebo-controlled study conducted in the United States. Subjects with a diagnosis of Dupuytren's contracture in a metacarpophalangeal (MP) or proximal interphalangeal (PIP) joint that resulted in a fixed flexion deformity of at least one finger, other than the thumb, that was at least 20° as measured by finger goniometry and was suitable for injection were randomized 2:1 to receive AA4500 0.58 mg or placebo.

This study was designed to be part of the larger clinical program, for adult patients with Dupuytren's contracture with a palpable cord, where the data from 2 pivotal Placebo-Controlled studies (AUX-CC-857 (NCT00528606) and AUX-CC-859 (NCT00533273)) and 7 non-pivotal studies were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of Dupuytren's contracture, with a fixed flexion deformity of at least one finger, other than the thumb, that had a contracture at least 20°, but not greater than 100°, for MP (80° for PIP) joints, caused by a palpable cord that had never been treated with AA4500.
* Had a positive "table top test," defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top.
* Judged to be in good health.

Exclusion Criteria:

* Had a chronic muscular, neurological, or neuromuscular disorder that affected the hands.
* Had received a treatment for Dupuytren's contracture, including surgery (fasciectomy or surgical fasciotomy), needle aponeurotomy/fasciotomy, or injection of verapamil and/or interferon on the selected primary joint within 90 days before the first dose of study drug.
* Had a known recent history of stroke, bleeding, a disease process that affected the hands, or other medical condition, which in the investigator's opinion, would make the subject unsuitable for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, Study Director — Endo Pharmaceuticals
Locations (15):
- United States (15):
  - 100 UCLA Medical Plaza, Suite 305, Los Angeles, California
  - Hand Surgery Clinic, Palo Alto, California
  - Hand Surgery Associates, PC, Denver, Colorado
  - The Hand and Upper Extremity Center of Georgia, P.C., Atlanta, Georgia
  - Rockford Orthopedic Associates, Ltd., Rockford, Illinois
  - The Indiana Hand Center, Indianapolis, Indiana
  - Brigham and Women's Hospital, Department of Orthopedic Surgery, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - TRIA Orthopaedic Center, Minneapolis, Minnesota
  - Hospital for Special Surgery, New York, New York
  - SUNY Stony Brook - Department of Orthopedics, Stony Brook, New York
  - Health Research Institute, Oklahoma City, Oklahoma
  - Hand Microsurgery & Reconstructive Orthopaedics, Erie, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Department of Orthopaedics, Brown University, Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Witthaut J, Bushmakin AG, Gerber RA, Cappelleri JC, Le Graverand-Gastineau MP. Determining clinically important changes in range of motion in patients with Dupuytren's Contracture: secondary analysis of the randomized, double-blind, placebo-controlled CORD I study. Clin Drug Investig. 2011 Nov 1;31(11):791-8. doi: 10.1007/BF03256918. PMID 21967070
- [Derived] Hurst LC, Badalamente MA, Hentz VR, Hotchkiss RN, Kaplan FT, Meals RA, Smith TM, Rodzvilla J; CORD I Study Group. Injectable collagenase clostridium histolyticum for Dupuytren's contracture. N Engl J Med. 2009 Sep 3;361(10):968-79. doi: 10.1056/NEJMoa0810866. PMID 19726771
- See also: XIAFLEX Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/125338lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.58 mg: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
- Placebo: Placebo injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
Period: Overall Study
Arm/Group | AA4500 0.58 mg | Placebo
Started | 204 | 104
Completed | 191 | 100
Not Completed | 13 | 4
Not completed — Withdrew consent | 4 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AA4500 0.58 mg | Placebo | Total
Number analyzed (Participants) | 204 | 104 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 57 | 177
  >=65 years | 84 | 47 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.7) | 63.3 (9.1) | 62.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 171 | 74 | 245
Race/Ethnicity, Customized [Number; unit: participants]
  White | 203 | 104 | 307
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 204 | 104 | 308

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success (Reduction in Contracture to 5° or Less) of the Primary Joint After the Last Injection
Description: The Primary Outcome Measure for patients treated with AA4500 is the percentage of joints that were successfully treated where "successfully treated" was defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
  The Primary Outcome Measure for placebo treated patients is the percentage of joints that were successfully treated where "successfully treated" was defined as reduction in contracture to within 0-5° of normal within 30 days of injection.
Time Frame: Within 30 days after the last injection
Population: Modified-Intent-to-Treat population (Intent-to-treat subjects were excluded from this population if they did not have fixed-flexion measurements after the first injection or had both screening and Treatment 1, Day 0 fixed-flexion measurements between 0 and 5 degrees)
Measure: Number; unit: Percentage of Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 203 | 103
Percentage of Joints | 64 | 6.8
Statistical Analysis 1: Comparison: AA4500 0.58 mg vs Placebo; p-value based on Cochran-Mantel-Haenszel test comparing treatment groups, stratified by baseline severity group and joint type; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Clinical Improvement After the Last Injection
Description: Clinical Improvement is defined as >= 50% reduction from baseline in degree of contracture within 30 days of the injection.
Time Frame: Baseline; within 30 days after the last injection
Population: Modified ITT population( Intent-to-treat subjects were excluded from this population if they did not have fixed-flexion measurements after the first injection or had both screening and Treatment 1, Day 0 fixed-flexion measurements between 0 and 5 degrees)
Measure: Number; unit: Percentage of Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 203 | 103
Percentage of Joints | 84.7 | 11.7

3. Secondary Outcome: Percent Reduction From Baseline Contracture After the Last Injection
Description: Percent change in degree of contracture measured as 100* (baseline contracture - last available post-injection contracture)/baseline contracture.
Time Frame: Baseline; within 30 days after the last injection
Population: Modified ITT population (Intent-to-treat subjects were excluded from this population if they did not have fixed-flexion measurements after the first injection or had both screening and Treatment 1, Day 0 fixed-flexion measurements between 0 and 5 degrees)
Measure: Mean (Standard Deviation); unit: Percent reduction from baseline
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 203 | 103
Percent reduction from baseline | 79.3 (32.58) | 8.6 (30.78)

4. Secondary Outcome: Change From Baseline Range of Motion After the Last Injection
Description: Change in degree of motion measured as last available post-injection range of motion - baseline range of motion.
Time Frame: Baselin; within 30 days after the last injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 198 | 103
degrees | 36.70 (21.01) | 4.0 (14.77)

5. Secondary Outcome: Time to First Achieve Success After the Last Injection
Time Frame: Last evaluation visit on which clinical success is achieved through the Day 30 evaluation
Population: Modified ITT population
Measure: Number; unit: percentage of joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 203 | 103
percentage of joints
  Injection 1, Day 1 | 12.8 | 0.0
  Injection 1, Day 7 | 12.3 | 0.0
  Injection 1, Day 30 | 14.3 | 1.0
  Injection 2, Day 0 | 0.5 | 0.0
  Injection 2, Day 1 | 4.9 | 0.0
  Injection 2, Day 7 | 5.4 | 0.0
  Injection 2, Day 30 | 6.4 | 1.0
  Injection 3, Day 0 | 0.0 | 0.0
  Injection 3, Day 1 | 2.0 | 0.0
  Injection 3, Day 7 | 2.5 | 0.0
  Injection 3, Day 30 | 2.5 | 4.9
  Day 90 | 0.5 | 0.0
  Did not reach clinical success by last injection | 36.0 | 93.2

6. Secondary Outcome: Clinical Success (Reduction in Contracture to 5° or Less) After the First Injection
Description: Clinical Success is defined as reduction in contracture to within 0-5 degrees of normal within 30 days of injection.
Time Frame: Within 30 days after first injection
Population: as for outcome 3
Measure: Number; unit: Percentage of Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 203 | 103
Percentage of Joints | 38.9 | 1.0

7. Secondary Outcome: Clinical Improvement After the First Injection
Description: Clinical Improvement is defined as >= 50% reduction from contracture within 30 days of the first injectionor greater of baseline contracture within 30 days of the injection.
Time Frame: Baseline; within 30 days after the first injection
Population: as for outcome 3
Measure: Number; unit: Percentage of Joints
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 203 | 103
Percentage of Joints | 67.5 | 2.9

8. Secondary Outcome: Percent Reduction From Baseline Contracture After the First Injection
Description: as for outcome 3
Time Frame: Baseline, within 30 days after the first injection
Population: Modified ITT population
Measure: Mean (Standard Deviation); unit: Percent reduction from baseline
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 203 | 103
Percent reduction from baseline | 64.8 (34.60) | 4.7 (20.81)

9. Secondary Outcome: Change From Baseline Range of Motion After the First Injection
Description: Change in degree of motion measured as last available post-injection range of motion - baseline range of motion.
Time Frame: Baseline; within 30 days after the first injection
Population: Modified ITT population (Change in degree of motion measured as last available post-injection range of motion - baseline range of motion)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500 0.58 mg | Placebo
Number analyzed (Participants) | 199 | 102
degrees | 28.30 (20.23) | 1.50 (11.03)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (non-SAEs) were collected from time of study drug administration, serious adverse events (SAEs) were collected from time subject signed ICF. Non-SAEs & SAEs were collected until 30 days after completion or discharge from study.
Description: This study was designed to be part of the larger clinical program. For information regarding XIAFLEX-associated Serious and Non-serious Adverse events please refer to the XIAFLEX Medication Guide & XIAFLEX Prescribing Information (see links above).
Arm/Group | AA4500 0.58 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/204 | 1/104
Other Adverse Events (participants affected / at risk) | 196/204 | 25/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=204) | Placebo (N=104)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.58 mg (N=204) | Placebo (N=104)
Blister (Skin and subcutaneous tissue disorders) | 11 (13) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 104 (178) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 51 (72) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 13 (16) | 0 (0)
Injection site haemorrhage (General disorders) | 76 (142) | 4 (4)
Injection site pain (General disorders) | 66 (117) | 5 (7)
Injection site pruritus (General disorders) | 11 (14) | 0 (0)
Injection site swelling (General disorders) | 43 (63) | 4 (4)
Lymph node pain (Blood and lymphatic system disorders) | 21 (25) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 20 (25) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 9 (9)
Oedema peripheral (General disorders) | 148 (296) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 65 (95) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (30) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 22 (25) | 0 (0)
Tenderness (General disorders) | 54 (85) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Auxilium Pharmaceuticals, Inc. agreements may vary with individual investigators but will not prohibit any investigator from publishing. Auxilium supports the publication of results from all centers of a multicenter trial but requests that reports based on single site data not preceed the primary publication of the entire clinical trial.